CLINICAL TRIAL: NCT02926950
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Added to Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo in Patients With Type 2 Diabetes Mellitus on Background of Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14834; 2016-001800-49 (EudraCT Number); U1111-1181-6145 (Other: UTN)
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin 400 mg + Metformin (Experimental): Following a 2-week run-in period, sotagliflozin 400 mg was administered as 2 tablets, once daily, before the first meal of the day plus metformin as prescribed by the Principal Investigator for up to 26 weeks in the double-blind Core Treatment Period, and participants continued the same treatment in the double-blind Extension Period for up to 53 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Metformin
- Placebo + Metformin (Placebo Comparator): Following a 2-week run-in period, matching placebo was administered as 2 tablets, once daily, before the first meal of the day plus metformin as prescribed by the Principal Investigator for up to 26 weeks in the double-blind Core Treatment Period, and participants continued the same treatment in the double-blind Extension Period for up to 53 weeks.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet. Route of administration: oral.
  Arms: Sotagliflozin 400 mg + Metformin
Drug: Placebo — Pharmaceutical form: tablet. Route of administration: oral.
  Arms: Placebo + Metformin
Drug: Metformin — Pharmaceutical form: tablet. Route of administration: oral.

SUMMARY:
Primary Objective:

To demonstrate the superiority of Sotagliflozin versus placebo on hemoglobin A1c (HbA1c) reduction in participants with type 2 diabetes (T2D) who have inadequate glycemic control with metformin.

Secondary Objectives:

* To compare Sotagliflozin versus placebo for.
* Change from baseline in 2-hour postprandial glucose (PPG) following a mixed meal.
* Change from baseline in fasting plasma glucose (FPG).
* Change from Baseline in systolic blood pressure (SBP) for participants with baseline SBP ≥130 millimeter of mercury (mmHg).
* Change from baseline in SBP for all participants.
* Change from baseline in body weight.
* Proportion of participants with HbA1c <6.5% and <7.0%.
* To evaluate the safety of Sotagliflozin versus placebo.

DETAILED DESCRIPTION:
The duration of the study period is up to 87 weeks, including a Screening Period consisting of a Screening phase of up to 2 weeks and a 2 week single blind Run-in phase, a 26 week double-blind Core Treatment Period, a 53-week double-blind Extension Period, a 4 week post treatment Follow-up period to collect safety information.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes currently treated with diet and exercise and on metformin at a stable dose ≥1500 milligrams per day (mg/day) for at least 12 weeks. However, participants on metformin at a dose <1500 mg/day at the time of enrollment (stable dose for at least 12 weeks before enrollment) may be eligible for screening if documentation of lack of tolerance of a metformin dose ≥1500 mg/day can be provided.
* Signed written informed consent.

Exclusion criteria:

* Age <18 years at Screening or < legal age of majority, whichever is greater.
* Type 1 diabetes mellitus.
* Body Mass Index (BMI) ≤20 or >45 kilograms per meter square (kg/m^2) at Screening
* Hemoglobin A1c <7% or >10% via central laboratory test at screening.
* Fasting plasma glucose (FPG) >15 millimole per liter (mmol/L) (270 milligrams per deciliter [mg/dL]) measured by the central laboratory at screening (Visit 1) and confirmed by a repeat test (>15 mmol/L [270 mg/dL]) before randomization.
* Women of childbearing potential not willing to use highly effective method(s) of birth control or who are unwilling or unable to be tested for pregnancy during the study.
* Treated with an antidiabetic pharmacological regimen other than metformin ≥1500 mg per day (or maximum tolerated dose) within the 12 weeks preceding the Screening Visit.
* Previous use of any types of insulin for >1 month (at any time, aside from pregnancy for treatment of gestational diabetes).
* History of prior gastric surgical procedure, including gastric banding, within 3 years before the Screening Visit.
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* Mean of 3 separate blood pressure measurements >180 mmHg (SBP) or >100 mmHg (diastolic blood pressure [DBP]).
* History of hypertensive urgency or emergency within 12 weeks prior to Screening.
* Participants with severe anemia, severe cardiovascular (including congestive heart failure New York Heart Association [NYHA] IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease or participants with short life expectancy making implementation of the protocol or interpretation of the study results difficult.
* Aspartate aminotransferase and/or alanine aminotransferase: >3 times the upper limit of the normal laboratory range.
* Total bilirubin: >1.5 times the upper limit of the normal laboratory range (except in case of Gilbert's syndrome).
* Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Participants who has taken other investigational drugs or prohibited therapy for this study within 12 weeks or 5 half-lives from screening or randomization, whichever is longer.
* Pregnant (confirmed by serum pregnancy test at Screening) or breastfeeding women.
* Participants is unwilling or unable to perform self-monitoring of blood glucose (SMBG), complete the participants diary, or comply with study visits and other study procedures as required per protocol.
* Contraindication to metformin as per local labelling.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (93):
- United States (67):
  - Investigational Site Number 8402003, Birmingham, Alabama
  - Investigational Site Number 8402017, Birmingham, Alabama
  - Investigational Site Number 8402052, Phoenix, Arizona
  - Investigational Site Number 8402056, Canoga Park, California
  - Investigational Site Number 8402020, Escondido, California
  - Investigational Site Number 8402028, Gold River, California
  - Investigational Site Number 8402067, Greenbrae, California
  - Investigational Site Number 8402025, Huntington Park, California
  - Investigational Site Number 8402051, La Mirada, California
  - Investigational Site Number 8402042, Lemon Grove, California
  - Investigational Site Number 8402011, Lincoln, California
  - Investigational Site Number 8402014, Long Beach, California
  - Investigational Site Number 8402066, Long Beach, California
  - Investigational Site Number 8402029, Los Angeles, California
  - Investigational Site Number 8402041, Los Angeles, California
  - Investigational Site Number 8402001, Los Angeles, California
  - Investigational Site Number 8402043, San Diego, California
  - Investigational Site Number 8402031, San Ramon, California
  - Investigational Site Number 8402047, Tarzana, California
  - Investigational Site Number 8402009, Boynton Beach, Florida
  - Investigational Site Number 8402016, Daytona Beach, Florida
  - Investigational Site Number 8402006, Hialeah, Florida
  - Investigational Site Number 8402035, Hialeah, Florida
  - Investigational Site Number 8402044, Hialeah, Florida
  - Investigational Site Number 8402045, Jacksonville, Florida
  - Investigational Site Number 8402026, Miami, Florida
  - Investigational Site Number 8402036, Miami, Florida
  - Investigational Site Number 8402064, Miami, Florida
  - Investigational Site Number 8402007, Miami, Florida
  - Investigational Site Number 8402061, Miami, Florida
  - Investigational Site Number 8402060, Miami Beach, Florida
  - Investigational Site Number 8402033, Opa-locka, Florida
  - Investigational Site Number 8402039, Orlando, Florida
  - Investigational Site Number 8402063, West Palm Beach, Florida
  - Investigational Site Number 8402038, Winter Haven, Florida
  - Investigational Site Number 8402008, Macon, Georgia
  - Investigational Site Number 8402054, Chicago, Illinois
  - Investigational Site Number 8402069, Newton, Iowa
  - Investigational Site Number 8402022, West Des Moines, Iowa
  - Investigational Site Number 8402059, Lexington, Kentucky
  - Investigational Site Number 8402068, Baton Rouge, Louisiana
  - Investigational Site Number 8402012, Metairie, Louisiana
  - Investigational Site Number 8402037, New Orleans, Louisiana
  - Investigational Site Number 8402053, New Orleans, Louisiana
  - Investigational Site Number 8402021, Rockville, Maryland
  - Investigational Site Number 8402062, Omaha, Nebraska
  - Investigational Site Number 8402005, Las Vegas, Nevada
  - Investigational Site Number 8402018, Greensboro, North Carolina
  - Investigational Site Number 8402002, Morehead City, North Carolina
  - Investigational Site Number 8402019, Oklahoma City, Oklahoma
  - Investigational Site Number 8402015, Eugene, Oregon
  - Investigational Site Number 8402058, Lansdale, Pennsylvania
  - Investigational Site Number 8402030, Dallas, Texas
  - Investigational Site Number 8402050, DeSoto, Texas
  - Investigational Site Number 8402010, Fort Worth, Texas
  - Investigational Site Number 8402040, Houston, Texas
  - Investigational Site Number 8402065, Houston, Texas
  - Investigational Site Number 8402057, Houston, Texas
  - Investigational Site Number 8402049, Magnolia, Texas
  - Investigational Site Number 8402046, Odessa, Texas
  - Investigational Site Number 8402013, San Antonio, Texas
  - Investigational Site Number 8402004, San Antonio, Texas
  - Investigational Site Number 8402023, Schertz, Texas
  - Investigational Site Number 8402027, Clinton, Utah
  - Investigational Site Number 8402032, Salt Lake City, Utah
  - Investigational Site Number 8402024, Virginia Beach, Virginia
  - Investigational Site Number 8402034, Seattle, Washington
- Canada (14):
  - Investigational Site Number 1242014, Barrie
  - Investigational Site Number 1242004, Brampton
  - Investigational Site Number 1242005, Brampton
  - Investigational Site Number 1242001, Concord
  - Investigational Site Number 1242007, Etobicoke
  - Investigational Site Number 1242010, Lévis
  - Investigational Site Number 1242012, Newmarket
  - Investigational Site Number 1242013, Oakville
  - Investigational Site Number 1242006, Pointe-Claire
  - Investigational Site Number 1242008, Sherbrooke
  - Investigational Site Number 1242015, Toronto
  - Investigational Site Number 1242002, Toronto
  - Investigational Site Number 1242003, Toronto
  - Investigational Site Number 1242011, Vancouver
- Hungary (6):
  - Investigational Site Number 3482002, Budapest
  - Investigational Site Number 3482003, Budapest
  - Investigational Site Number 3482006, Budapest
  - Investigational Site Number 3482004, Debrecen
  - Investigational Site Number 3482001, Esztergom
  - Investigational Site Number 3482007, Nyíregyháza
- Slovakia (6):
  - Investigational Site Number 7032001, Bratislava
  - Investigational Site Number 7032005, Bratislava
  - Investigational Site Number 7032003, Malacky
  - Investigational Site Number 7032002, Nitra
  - Investigational Site Number 7032004, Štúrovo
  - Investigational Site Number 7032006, Trenčín

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and supporting clinical documents are available for request at clinicalstudydatarequest.com. While making information available we continue to protect the privacy of the participants in our clinical trials and to remove commercially confidential information (CCI). Details on Data Sharing criteria and process for requesting access can be found at this web address: clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 87 investigative sites in Canada, Hungary, Slovakia and the United States from 11 November 2016 to 22 March 2019.
Pre-assignment Details: Participants with a diagnosis of type 2 Diabetes Mellitus were enrolled in 1 of 2 treatment groups, Sotagliflozin 400 milligrams (mg) once daily (QD) + Metformin and Placebo + Metformin. Participants were randomly assigned to the ratio of 1:1 to these reporting groups.
Groups:
- Placebo + Metformin: Following a 2-week run-in period, matching placebo was administered as 2 tablets, QD, before the first meal of the day plus Metformin as prescribed by the Principal Investigator for up to 26 weeks in the double-blind Core Treatment Period, and participants continued the same treatment in the double-blind Extension Period for up to 53 weeks.
- Sotagliflozin 400 mg + Metformin: Following a 2-week run-in period, Sotagliflozin 400 mg was administered as 2 tablets, QD, before the first meal of the day plus Metformin as prescribed by the Principal Investigator for up to 26 weeks in the double-blind Core Treatment Period, and participants continued the same treatment in the double-blind Extension Period for up to 53 weeks.
Period: Overall Study
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Started | 259 | 259
Completed | 210 | 211
Not Completed | 49 | 48
Not completed — Adverse Event | 4 | 6
Not completed — At the participant's own request | 21 | 25
Not completed — Reason not Specified | 17 | 9
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin | Total
Number analyzed (Participants) | 259 | 259 | 518
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.4) | 60.0 (10.1) | 59.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 117 | 230
  Male | 146 | 142 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106 | 117 | 223
  Not Hispanic or Latino | 153 | 140 | 293
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 19 | 6 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 40 | 28 | 68
  White | 197 | 223 | 420
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.19 (0.82) | 8.20 (0.78) | 8.20 (0.80)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 133.80 (13.95) | 134.06 (13.95) | 133.93 (13.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline and Week 26
Population: Intent-to-treat (ITT) population included all randomized participants. Missing data was imputed using the retrieved dropouts and washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
percentage of HbA1c | -0.29 (0.079) | -0.77 (0.077)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 26 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares (LS) Means = -0.47, 95% CI 2-sided [-0.64 to -0.309], Standard Error of Mean 0.084

2. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following a Mixed Meal at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 26
Population: ITT population included all randomized participants. Missing data are imputed using control-based copy reference multiple imputation method.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
millimole per liter (mmol/L) | -0.930 (0.2353) | -2.502 (0.2292)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and country as fixed effects, and baseline 2- hour postprandial glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.572, 95% CI 2-sided [-2.0538 to -1.0909], Standard Error of Mean 0.2457

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 26
Population: ITT population included all randomized participants. Missing data was imputed using the retrieved dropouts and washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
mmol/L | -0.550 (0.1864) | -1.310 (0.2089)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 26 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline fasting plasma glucose as a covariate; Test type: Superiority; p = 0.0007, ANCOVA; Difference in LS Means = -0.76, 95% CI 2-sided [-1.2006 to -0.3198], Standard Error of Mean 0.2247

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
kilogram (kg) | -0.69 (0.310) | -2.56 (0.331)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 26 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and country as fixed effects, and baseline weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.87, 95% CI 2-sided [-2.591 to -1.144], Standard Error of Mean 0.369

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 12 in Participants With Baseline SBP ≥130 mmHg
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 12
Population: Analysis was performed on ITT population in participant with baseline SBP ≥130 mmHg. Missing data was imputed using control-based copy reference multiple imputation method.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 129 | 137
millimeter of mercury (mmHg) | -6.92 (1.233) | -10.21 (1.270)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 12 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤ 8.0, >8.0%) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.0209, ANCOVA; Difference in LS Means = -3.28, 95% CI 2-sided [-6.07 to -0.497], Standard Error of Mean 1.422

6. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 12
Population: ITT population included all randomized participants. Missing data was imputed using control-based copy reference multiple imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
mmHg | -1.87 (0.949) | -5.41 (0.950)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; The change from baseline to Week 12 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤ 8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.0004, ANCOVA; Difference in LS Means = -3.54, 95% CI 2-sided [-5.479 to -1.592], Standard Error of Mean 0.992

7. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
percentage of participants | 5.4 | 10.8
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; Percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening. Missing data at Week 26 were assigned a status of nonresponder in the analysis; Test type: Superiority; p = 0.0238, Cochran-Mantel-Haenszel; Percentage Difference = 5.4, 95% CI 2-sided [0.75 to 10.06]

8. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
percentage of participants | 15.8 | 29.7
Statistical Analysis 1: Comparison: Placebo + Metformin vs Sotagliflozin 400 mg + Metformin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Percentage Difference = 13.9, 95% CI 2-sided [6.91 to 20.89]

9. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤70 mg/dL]. Participants may be reported in more than one category.
Time Frame: Up to 79 weeks in the treatment period
Population: Safety population was defined as all randomized participants who had received at least 1 dose of the double-blind investigational medicinal product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
Number analyzed (Participants) | 259 | 259
percentage of participants
  Any hypoglycemia | 11.6 | 6.6
  Documented symptomatic hypoglycemia | 6.2 | 3.1
  Severe or documented symptomatic hypoglycemia | 6.2 | 3.1

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 79 weeks) + 4 weeks
Description: Safety population was defined as all randomized participants who had received at least 1 dose of the double-blind investigational medicinal product (IMP). Hypoglycemia was captured and handled separately from other adverse events and is reported in the outcome measure section.
Arm/Group | Placebo + Metformin | Sotagliflozin 400 mg + Metformin
All-Cause Mortality (participants affected / at risk) | 1/259 | 3/259
Serious Adverse Events (participants affected / at risk) | 23/259 | 19/259
Other Adverse Events (participants affected / at risk) | 109/259 | 85/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin (N=259) | Sotagliflozin 400 mg + Metformin (N=259)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral artery thrombosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin (N=259) | Sotagliflozin 400 mg + Metformin (N=259)
Hypertension (Vascular disorders) | 13 | 3
Headache (Nervous system disorders) | 15 | 6
Diarrhoea (Gastrointestinal disorders) | 11 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 8
Vitamin D deficiency (Metabolism and nutrition disorders) | 19 | 14
Bronchitis (Infections and infestations) | 17 | 5
Nasopharyngitis (Infections and infestations) | 17 | 14
Upper respiratory tract infection (Infections and infestations) | 20 | 20
Urinary tract infection (Infections and infestations) | 15 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT02926950/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT02926950/SAP_001.pdf